CLINICAL TRIAL: NCT02561624
Title: Expanding the Successful E-voucher System to Improve Malaria Prevention and Fight New Global Health Threats Through Innovative Health Partnerships and Mobile Phone Technology in Tanzania
Brief Title: Hati Salama (Secure Voucher)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Mennonite Economic Development Associates (Unknown)
Responsible Party: Principal Investigator, Dr. Karen Yeates, Associate Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DMED-1712-14
Record Dates: First submitted 2015-07-20; First posted 2015-09-28 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Malaria
Keywords: mHealth; Text message
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Use of behaviour change communication via text messages to pregnant women receiving an electronic voucher for long lasting insecticide treated nets redemption through antenatal clinics.
  Interventions: Behavioral: Behaviour change communication via text message
- Control (No Intervention): Control group receives no behaviour change communication via text message, but receives an electronic voucher for long lasting insecticide treated nets redemption through antenatal clinics.

INTERVENTIONS:
Behavioral: Behaviour change communication via text message
  Arms: Intervention

SUMMARY:
The use of long-lasting insecticide treated nets (LLINs) is shown to reduce malaria prevalence. The Tanzania Net Voucher Scheme has been an active component of bed net distribution to pregnant women in Tanzania since 2004. The transition from paper vouchers to electronic vouchers in this program has increased efficiency and the ability to track and distribute nets since 2007. Although the program has been successful, to date, electronic voucher redemption varies widely across the country and it has not been clearly established as to what barriers exist for women who receive electronic vouchers in the program. This cluster-randomized trial was designed to examine perceived barriers to electronic voucher redemption among pregnant women and to evaluate if educational and personalized text messages around electronic voucher redemption and bed net usage will increase electronic voucher redemption when directed at pregnant women who receive electronic vouchers in the currently existing program.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women capable of providing informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5219 (Actual)
Dates: Start 2015-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Increased uptake of long-lasting insecticide treated nets from retailers using an electronic voucher through text messaging. | 12 weeks
  The outcome measure will be assessed by LLIN evoucher redemption.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Yeates, MD, Principal Investigator — Queen's University
Locations (1):
- Pamoja Tunawez, Moshi, Tanzania

REFERENCES:
- [Derived] Vey T, Kinnicutt E, Day AG, West N, Sleeth J, Nchimbi KB, Yeates K. Targeted Behavior Change Communication Using a Mobile Health Platform to Increase Uptake of Long-Lasting Insecticidal Nets Among Pregnant Women in Tanzania: Hati Salama "Secure Voucher" Study Cluster Randomized Controlled Trial. J Med Internet Res. 2025 Mar 19;27:e51524. doi: 10.2196/51524. PMID 40106816
- [Derived] Vey T, Kinnicutt E, West N, Sleeth J, Nchimbi KB, Yeates K. Implementation of a Mobile Health Approach to a Long-Lasting Insecticidal Net Uptake Intervention for Malaria Prevention Among Pregnant Women in Tanzania: Process Evaluation of the Hati Salama (HASA) Randomized Controlled Trial Study. J Med Internet Res. 2024 Nov 5;26:e51527. doi: 10.2196/51527. PMID 39499551